CLINICAL TRIAL: NCT02859675
Title: Olfactogustatory Perception, Eating Behaviour and Inflammation in Crohn's Disease
Acronym: Smell&Crohn
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BRONDEL Ass INRA 2011
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Crohn's Disease; Olfactogustatory Perception
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Crohn and anti-TNF treatment: Tests at 3 or 4 weeks after the beginning of anti-TNF treatment
  Interventions: Other: triangular test; Biological: blood sampling; Other: Questionnaires
- Crohn and without anti-TNF treatment: tests performed according to patient availability
  Interventions: Other: triangular test; Biological: blood sampling; Other: Questionnaires
- Control: tests performed according to patient availability
  Interventions: Other: triangular test; Biological: blood sampling; Other: Questionnaires

INTERVENTIONS:
Other: triangular test — metabolic state, impedance measurement, potential flavours evoked by sucrose,
Biological: blood sampling — sampling of 2 mL
Other: Questionnaires — Stunkard, PrefQuest

SUMMARY:
This study will improve our understanding of the mechanisms underlying anorexia in persons with Crohn's disease flare-ups. The practical spin-off from this research is potentially very important for the management of nutritional disorders associated with the disease by guiding diets towards foods that correspond to patients' preferences and/or to modified tastes. In addition, the results could lead to the identification of sensory markers that herald an inflammatory flare-up of the disease.

ELIGIBILITY:
For patients :

Inclusion Criteria:

* Age between 18 and 60 years,
* Diagnosis of Crohn's disease according to clinical, endoscopic, histological, radiological and biochemical criteria as defined by the European Consensus Conference,
* Men or women who have provided consent and willing to cooperate.

Exclusion Criteria:

* Chronic inflammatory intestinal disease (CIID) other than Crohn's disease: haemorrhagic rectocolitis, undetermined colitis, microscopic colitis.
* Intercurrent disease (diabetes and metabolic disease, liver cirrhosis, progressive cancer, acute or chronic infection, Human Immunodeficiency Virus HIV),
* Organ failure (respiratory, heart, or renal failure, neurological disorders),
* Intolerance to gluten,
* Treatments (other than those used for Crohn's disease) able to interfere with food intake,
* Aversion to foods consumed or smelled,
* Poor understanding of cognitive tasks required.
* Crohn's disease complicated by an abscess or infectious complication
* Acute Crohn's disease defined by a CDAI score > 150

For Controls:

Inclusion Criteria:

* Adult person
* Without follow-up for a chronic pathology
* Having given its consent

Exclusion Criteria:

* Protected adult
* Person not affiliated to a social security system
* Pregnant or breastfeeding woman
* Active smoker
* No one who does not speak French
* Taking treatment that interferes with taste or acts on the central nervous system

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: understanding of the mechanisms underlying anorexia in persons with Crohn's disease flare-ups
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Modification of sweet taste | through the study completion up to 10 years
  the measurement of detection thresholds consists in presenting to the participants in order of increasing concentrations, series of forced-choice triangular tests

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France